CLINICAL TRIAL: NCT04577482
Title: Real World Evidence of the Effectiveness and Clinical Practice Use of Glecaprevir/Pibrentasvir in DAA Treatment-Experienced Patients With Chronic Hepatitis C Genotype 1 in Russian Federation (CHOICE)
Brief Title: Study of Oral Glecaprevir/Pibrentasvir Tablets in Participants Aged 12 Years or Older With Chronic Hepatitis C to Assess Sustained Virological Response
Acronym: CHOICE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-397
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Hepatitis C Virus (HCV); Chronic Hepatitis C Infection; Glecaprevir/pibrentasvir; GLE/PIB; CHOICE; Chronic Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants treated with Glecaprevir/Pibrentasvir: Participants will receive glecaprevir/pibrentasvir (GLE/PIB) as prescribed by physician in accordance with local clinical practice.

SUMMARY:
Hepatitis C virus (HCV) infection is among the most common of all chronic liver diseases. HCV predominantly affects liver cells and causes the liver to become inflamed and damaged. This can lead to cirrhosis (scarring of the liver), liver cancer or the need for liver transplant. This study will evaluate how effective glecaprevir/pibrentasvir (GLE/PIB) is in participants with chronic HCV infection. Effectiveness will be assessed as the achievement of sustained virologic response.

GLE/PIB is an approved drug for the treatment of HCV. Participants 12 years or older with chronic HCV infection will be enrolled. This is a prospective (conducted in future) study in therapy of direct-acting antiviral (DAA) treatment-experienced participants with chronic hepatitis C genotype 1. Around 67 participants will be enrolled at multiple sites in Russian Federation.

Participants will receive oral GLE/PIB tablets as prescribed by the physician in accordance with local clinical practice, international guidelines and/or label. Prescription is independent from this study and is decided before providing opportunity to the participate in the study.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice and participants will be followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Direct-acting antiviral treatment-experienced participants with confirmed chronic hepatitis C (CHC) genotype 1, receiving combination therapy with the all oral glecaprevir/pibrentasvir (GLE/PIB) regimens according to standard of care, international guidelines and in line with the current local label.
* Participants can enroll up to 4 weeks after starting treatment

Exclusion Criteria:

- Participating or intending to participate in a concurrent interventional therapeutic trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with hepatitis C virus (HCV) infection of genotype 1 prescribed with glecaprevir/pibrentasvir in accordance with local clinical practice and label.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Sustained Virological Response (SVR) at Week 12 (SVR12) | Week 12 after the end of treatment
  SVR12 is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) < 50 IU/ml or lower limit of quantification/detection (LLoQ/D) available at the site at Week 12 after the last actual dose.

SECONDARY OUTCOMES:
Percentage of Participants Achieving SVR12 | Week 12 after the end of treatment
  SVR12 is defined as HCV RNA < LLoQ/D 12 weeks after the last actual dose of GLE/PIB with a sensitive polymerase chain reaction (PCR) available in the clinical site in the settings of the Russian Federation in subgroups of interest.
Number of Participants With Co-morbidities and Taking Concomitant Medication | Up to Week 12 after the end of treatment
  Number of participants with co-morbidities and taking concomitant medication of interest report will be calculated.
Health Care Resource Utilization (HCRU) | Up to Week 12 after the end of treatment
  HCRU will be total number of visits/touchpoints (face to face or phone call) with a Health Care Provider (HCP) or designee in relation to their HCV infection during the study as recorded overall and by subpopulations of interest.
Percent of Glecaprevir/Pibrentasvir Dose Taken by Participant Report in Relation to the Prescribed Target Dose | Up to Week 12 after the end of treatment
  Number of pills taken out of the number that should have been taken will be calculated.
Number of Participants With Adverse Events (AEs) | Up to Week 12 after the end of treatment
  An adverse event (AE) is defined as any untoward medical occurrence in a patient which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug overall and in subgroups of interest. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Percentage of Participants Who Experienced Post-Baseline Shifts in Clinical Laboratory Values | Up to Week 12 after the end of treatment
  Percentage of participants who experience post-baseline shifts during treatment in clinical laboratory values will be summarized overall and in subgroups of interest.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- Russia (10):
  - South Ural State Medical University /ID# 226555, Chelyabinsk
  - LLC Center of Targeted Therapy /ID# 239529, Domodedovo
  - Irkutsk Regional Center for the Prevention and Control of AIDS and Infections /ID# 229509, Irkutsk
  - Specialized Clinical Infectious Diseases Hospital /ID# 229814, Krasnodar
  - Infectious Clinical Hosp #1 /ID# 225063, Moscow
  - Infectious Clinical Hospita l#2 /ID# 243217, Nizhny Novgorod
  - S. P. Botkin City Hospital /ID# 229510, Oryol
  - Saint-Petersburg AIDS Center /ID# 239357, Saint Petersburg
  - Samara Region Clinical HIV/AIDS Prevention and Control Center /ID# 226591, Samara
  - Stavropol State Medical University /ID# 243216, Stavropol

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-397#additional-resources-section